CLINICAL TRIAL: NCT07165756
Title: "Mon Parcours de Vie" Localized Breast Cancer: Announcement, Support, Information on the Disease and Treatments. Pilot Study to Assess the Value of Written Information Documents.
Acronym: MaVie
Status: Recruiting | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A00330-49
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-05

CONDITIONS: Localized Breast Cancer
Keywords: Announcement of cancer and treatment; Breast cancer; Information documents
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since late 2019, the French association "MON PARCOURS DE VIE" has developed books donated by caregivers at cancer centers in France. These documents are available online: https://www.monparcoursdevie.fr/. They are highly acclaimed by women suffering from the breast cancer, as well as by caregivers. Four volumes have been written: 'Metastatic breast cancer', 'Localized breast cancer', 'Preserving my well-being', 'After breast cancer', and finally 'Breast cancer, support and accompaniment'.

The aim in writing these information brochures is to provide clear, concise, useful information, with pedagogy, gentleness, benevolence, humility, cheerfulness, imagination, simplicity and an innovative presentation. These documents are a new and innovative method of providing information, delivered by caregivers who work with women suffering from breast cancer. It extends the human support so necessary in this disease.

It seemed important to us to evaluate, through a clinical study, the impact of the written documents "Mon Parcours de Vie" - volume 2: Breast cancer and volume 3: Preserving my well-being, concerning the announcement of a localized breast cancer in the initial management for the first time in the breast pathway. The objectives of the clinical study are to evaluate the acceptability and impact of these two written information documents on anxiety generated by the announcement of cancer and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with localized breast cancer consulting for medical treatment (chemotherapy+/- immunotherapy+/anti-HER2 targeted therapy)
* Diagnosis of invasive breast cancer for which there is an indication for local and medical treatment.
* WHO ≤ 1
* Patient has understood, signed and dated the consent form
* Patient affiliated to the social security system

Exclusion Criteria:

* Patient with metastatic breast cancer
* History of other cancer
* Patient unable to read or speak French
* Persons deprived of liberty or under guardianship (including curatorship).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected based on the scheduling of a medical consultation for the announcement of medical treatments (chemotherapy+/- immunotherapy+/anti-HER2 targeted therapy) for breast cancer at our Institute.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability rate | 14 days
  Acceptability rate will be measured by the proportion of patients who accepted and read in full the 2 documents distributed; comparison of acceptability between the two information documents.
Variation in the anxiety score | 14 days
  Variation in the anxiety score will be assessed by the anxiety score established from questions relating to anxiety on the Hospital Anxiety and Depression Scale (HADS) at the consultation for the announcement of medical treatments (chemotherapy+/- immunotherapy+/anti-HER2 targeted therapy) with the distribution of written documents (=D0) and immediately after reading the documents (max at D14 after inclusion).

SECONDARY OUTCOMES:
Level of understanding | 14 days
  After reading the documents, the level of understanding will be assessed for the period of cancer diagnosis, treatment and preservation of well-being.
Audience of documents | 14 days
  The audience of the documents will be assessed by the patient's interest in the documents and her expectations (interest in volume 2 and volume 3 (interested in both); also possible comparison of the audience between the two documents.
Perception and comprehension of the documents | 14 days
  Perception and comprehension of the documents will be determined by assessing readability, perception of information and presentation.
Patient's level of satisfaction | 14 days
  The patient's level of satisfaction with the documents will be measured by the evaluation questionnaire (satisfaction score for each of the two volumes).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France